CLINICAL TRIAL: NCT04455243
Title: Pilot Double Blinded Randomized Placebo Controlled Multi Central Clinical Trial on Inflammatory Regulation Effect of NAC on COVID-19
Brief Title: Inflammatory Regulation Effect of NAC on COVID-19 Treatment
Acronym: INFECT-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Tariq Alhawassi (Other)
Responsible Party: Sponsor-Investigator, Dr. Tariq Alhawassi, Chairman of Clinical Trial Support Unit, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-20-4934
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: NAC
MeSH Terms: conditions — COVID-19 | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: N-Acetyl cysteine
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetyl cysteine — 150 mg/kg every 12 hours for 14 days (oral/IV) Diluted in 200 ml diluent (D5%, NS)
  Other Names: NAC
  Arms: Intervention group
Drug: Placebo — Matching placebo administered in the same schedule and volume as NAC
  Arms: Control group

SUMMARY:
Study times to evaluate the efficacy of N-Acetylcysteine therapy in the management of adult admitted patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult above 18 years of age
* Admitted to the hospital With confirmed COVID-19 by RT-PCR test
* On oxygen supplement

Exclusion Criteria:

* Active use of NAC
* Known NAC allergy
* In the opinion of the treating team, progression of death is imminent and inevitable within the next 24 hour, irrespective of provision treatment
* All patients enrolled in any other investigational drug studies in COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to Recovery | 28 days
  Day of recovery is defined as the first day on which of the following three categories from The Ordinal Scale on Covid-19 Clinical Improvement
  1. Not-Hospitalized, No limitation on activity.
  2. Not Hospitalized, with limitation on activity.
  3. Hospitalized, Not requiring supplemental Oxygen

IPD SHARING:
Plan to Share IPD: Undecided
IPD data will be shared. However, the exact sharing plans on what or when is not yet decided.